CLINICAL TRIAL: NCT06411249
Title: A Phase 4, Multicenter, Prospective, Open-Label Study Describing the Efficacy and Safety of Belimumab Administered Subcutaneously in Adult Participants With Early Systemic Lupus Erythematosus
Brief Title: A Study Describing the Efficacy and Safety of Belimumab Administered in Adult Participants With Early Systemic Lupus Erythematosus (SLE)
Acronym: BE-EARLY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 219240; 2023-509146-35-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Belimumab; Benlysta; Efficacy; Safety; Early Use; Systemic Lupus Erythematosus; Autoimmune Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belimumab (GSK1550188) (Experimental): Participants will receive GSK1550188.
  Interventions: Drug: Belimumab (GSK1550188)

INTERVENTIONS:
Drug: Belimumab (GSK1550188) — GSK1550188 will be administered subcutaneously.
  Other Names: BEL (BENLYSTA)

SUMMARY:
This is a prospective, open-label, single arm 3-year clinical study to describe the short-term and long-term efficacy and safety of belimumab in participants with autoantibody positive early SLE with ongoing disease activity despite stable initial SLE therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of systemic lupus erythematosus (SLE) within 2 years of signing the informed consent according to the European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) SLE classification criteria 2019
* Have unequivocally positive autoantibody test results defined as an Anti-nuclear antibody (ANA) titer greater than or equal to (≥) 1:80 and/or a positive anti-Double stranded deoxyribonucleic acid (dsDNA) serum antibody test from 2 independent time points
* Active SLE defined as:
* Clinical SLEDAI-2K (excluding anti-dsDNA and C3/C4) score greater than (>) 4, OR
* Clinical SLEDAI-2K (excluding anti-dsDNA and C3/C4) less than or equal to (≤) 4 and prednisone or equivalent dose ≥10 milligram per day (mg/day)
* The Systematic Lupus International Collaborating Clinics/American College of Rheumatology (SLICC/ACR) Damage Index (SDI) = 0 at Screening
* Male and/or female; a female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* Not a Woman of childbearing potential (WOCBP) OR
* Is a WOCBP and using a contraceptive method that is highly effective
* Capable of giving signed informed consent

Exclusion criteria:

* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to SLE (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal (GI), hepatic, renal, neurological, psychiatric, malignancy, or infectious diseases) and/or a planned surgical procedure, which, in the opinion of the principal investigator (PI), could confound the results of the clinical study or put the participant at undue risk.
* Participants with history of major organ transplant or hematopoietic stem cell/marrow transplant or renal transplant.
* Have an acute or chronic infection including requiring management as follows:
* Currently on any suppressive therapy for a chronic infection such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria.
* A serious infection requiring treatment with intravenous or Intramuscular (IV/IM) antibiotics and/or hospitalization if the last dose of antibiotics or the hospital discharge date was within 60 days of the first day of dosing (Day 1). Prophylactic anti-infective treatment is allowed.
* Confirmed active or untreated latent tuberculosis (TB):
* Diagnosis of active TB confirmed by: 1) evidence of active TB disease from chest imaging (posterior anterior and lateral x-rays or chest computed tomography [CT]), 2) medical history and physical examination, and 3) either positive microscopy smear/culture for mycobacteria or positive TB polymerase chain reaction (PCR), i.e., Xpert. A tuberculin skin test (TST) or an interferon gamma release assay (IGRA) will be done for all participants. A positive TST or a positive (not indeterminate) IGRA TB test such as QuantiFERON-TB Gold Plus test is indicative but not required for diagnosis of active TB. A positive TST is defined as a skin induration ≥5 millimeter (mm) at 48 to 72 hours (regardless of Bacillus Calmette-Guerin or other vaccination history).
* Untreated latent tuberculosis infection (LTBI) confirmed by: 1) no evidence of active TB based on chest imaging, medical history and physical examination and laboratory evaluation of sputum; and 2) a positive TST, defined as a skin induration >5 mm at 48 to 72 hours, regardless of Bacillus Calmette-Guerin or other vaccination history); or a positive (not indeterminate) IGRA TB test such as QuantiFERON-TB Gold Plus test. Those with IGRA positive tests or positive TST who can document ongoing LTBI treatment for at least 4 weeks may be enrolled. Those with IGRA positive tests with documentation of the following may also be enrolled:
* Successful completion of treatment for active TB.
* Completion of treatment for LTBI (with treatment as per local practice, for example: 3 months of isoniazid and rifampin or 4 months of rifampin or 3 months weekly isoniazid and rifapentine, or 9 months of isoniazid).
* Confirmed Progressive multifocal leukoencephalopathy (PML) or unexplained new-onset or deteriorating neurologic signs and symptoms.
* Have severe active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, Cerebrovascular accident (CVA), cerebritis, or CNS vasculitis) requiring therapeutic intervention within 60 days of Screening.
* Active Lupus Nephritis defined as active urinary sediment and/or proteinuria >500 milligrams (mg) per 24 hours, or equivalent using spot urine protein to creatinine ratio, requiring induction therapy not permitted by protocol.
* Participants with patient health questionnaire (PHQ)-9 score ≥10 that in the opinion of a mental healthcare professional pose a serious suicide risk, or any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months, or who in the investigator's judgment, poses a significant suicide risk. NOTE: For participants with a PHQ-9 score ≥10, at the Screening visit or at the day 1 visit before the first administration of the study drug, it is required that they be referred for an assessment by a mental healthcare professional (e.g., locally licensed psychiatrist, psychologist, or master's level therapist) before the investigator makes a final decision regarding suitability for enrollment.
* Known to have titers of human anti-mouse antibody or history of hypersensitivity reactions when treated with diagnostic or therapeutic monoclonal antibodies
* Live or live-attenuated vaccine(s) within 35 days prior to Screening or plans to receive such vaccines during the Screening period or during the clinical study
* Chronic oral steroid use for a non-SLE disorder at the Screening study visit (e.g., for asthma). Inhaled steroid use will be allowed.
* Treatment at or prior to Screening study visit:
* Treatment at Screening study visit with any of the following:
* Azathioprine (AZA) >200 mg/day
* Methotrexate (MTX) (any formulation) >25 mg/week
* Mycophenolate mofetil (MMF) (oral [PO])/MMF hydrochloride (IV) >2 grams (g)/day
* Mycophenolate acid/sodium (PO) >1.44 g/day
* Oral cyclophosphamide >2.5 mg/kilograms (kg)/day
* Tacrolimus >0.2 mg/kg/day
* Cyclosporine (PO) >2.5 mg/kg/day
* Treatment within specified timeframe prior to Screening:
* Intra-articular, IM, or IV corticosteroids within 6 weeks of Day 1
* Daily use of >1 Nonsteroidal anti-inflammatory (NSAID) within 2 weeks prior to Day 1
* Treatment at any time prior to Screening with any of the following:
* Second line use of conventional immunosuppressants (ISs) or anti-malarials (AMs)
* Commercially available Belimumab (BEL)
* Anifrolumab
* Rituximab or other B cell depleting therapies
* Anti-tumor necrosis factor (TNF) therapy (e.g., adalimumab, etanercept, infliximab)
* Other treatments with effects on the immune system (e.g., abatacept, interleukin-1 receptor antagonist [anakinra], Janus kinase (JAK) inhibitors)
* IV cyclophosphamide
* IV immunoglobulin
* Plasmapheresis
* History of primary immunodeficiency, or hypogammaglobulinemia (Immunoglobulin G [IgG] <400 mg/deciliter [dL]) or Immunoglobulin A (IgA) deficiency (IgA <10 mg/dL) at Screening
* Have a Grade 3 or greater neutropenia, defined as absolute neutrophil count <1000/cubic millimeter (mm3) (<1.0 x109/liter [L]) based on the Common terminology criteria for adverse events (CTCAE) version (v) 5.0
* Alanine aminotransferase >2 x upper limit of normal (ULN)
* Total bilirubin >1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]). Participants with Gilbert's syndrome can be included with total bilirubin >1.5xULN as long as direct bilirubin is ≤1.5xULN. Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice. NOTE: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome), asymptomatic gallstones, and chronic stable hepatitis B (in whom Hepatitis D [HDV] has been excluded) or C are acceptable if participant otherwise meets entry criteria.
* Have any other clinically significant abnormal laboratory value, that in the opinion of the investigator, is capable of significantly altering the absorption, metabolism, or elimination of the clinical study intervention; or constitutes a risk when taking the clinical study intervention or interferes with the interpretation of the clinical study data.
* Positive Human immunodeficiency virus (HIV) antibody test
* Serologic evidence of Hepatitis B (HB) infection based on the results of testing for hepatitis B surface antigen (HBsAg), anti-hepatitis B core (HBc) and anti-HBs will be excluded as follows:
* Participants positive for HBsAg.
* Participants negative for HBsAg but positive for Anti-HBc and detectable hepatitis B virus (HBV) DNA, regardless of Anti-HBs antibody status.
* Positive Hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention. NOTE: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C Ribonucleic acid (RNA) test is obtained.
* Positive Hepatitis C RNA test result at Screening or within 3 months prior to first dose of study intervention. NOTE: Test is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.
* Sensitivity to the clinical study intervention, or components thereof, or monoclonal antibodies or drug or other allergy that, in the opinion of the investigator, contraindicates participation in the clinical study
* Current drug or alcohol dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 1
* Current enrolment or past participation in any other clinical study involving an investigational study intervention (including investigational vaccines) within 3 months or 5 half-lives of the investigational drug (whichever is longer) before enrolment
* Unable to administer clinical study intervention by subcutaneous (SC) auto-injector at home and has no other reliable resource to administer the study intervention at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-05-29 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of Participants Achieving Lupus Low Disease Activity State (LLDAS) at Week 52 | At Week 52
  LLDAS is defined as Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) less than or equal to (≤) 4, with no activity in major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, fever) and no new features of lupus disease activity compared with the previous assessment, Physician Global Assessment (PGA) ≤ 1, with a 7-day average oral prednisone equivalent dose for SLE reasons ≤7.5 milligram (mg)/day and stable treatment and without discontinuing due to lack of efficacy, dying, or taking prohibited medications.

SECONDARY OUTCOMES:
Part A: Percentage of Participants Achieving SLE Responder Index 4 (SRI4) at Week 52 | At Week 52
  SRI4 is defined as greater than or equal to (≥) 4-point reduction from baseline in SLEDAI-2K score and no worsening (increase of < 0.30 points from baseline) in PGA and no new Easy- British Isles Lupus Assessment Group (BILAG) A organ domain score or 2 new Easy-BILAG B organ domain scores compared with baseline at the time of assessment without participants discontinuing due to lack of efficacy, dying, taking prohibited medications or meeting treatment failure criteria.
Part A: Percentage of Participants Achieving Lupus Low Disease Activity State (LLDAS) for ≥ 25 percent (%) of time from Day 1 to Week 52 | Day 1 and up to Week 52
  LLDAS is defined as Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) less than or equal to (≤) 4, with no activity in major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, fever) and no new features of lupus disease activity compared with the previous assessment, Physician Global Assessment (PGA) ≤ 1, with a 7-day average oral prednisone equivalent dose for SLE reasons ≤7.5 milligram (mg)/day and stable treatment and without discontinuing due to lack of efficacy, dying, or taking prohibited medications.
Part A: Percentage of Participants Achieving Average Oral Prednisone Equivalent Dose ≤ 5 mg/day at Week 52 | At Week 52
  A seven-day average oral prednisone equivalent dose ≤5 mg/day at week 52, if oral prednisone equivalent dose is >5 mg/day at baseline without study intervention discontinuation due to lack of efficacy, serious AE, prohibited medication intake, or treatment failure by Week 52.
Part A: Estimate of probability of having a Severe Flare defined as modified SELENA-SLEDAI Flare Index (SFI) at Week 52 | At Week 52
  SFI Flare was defined as a mild/moderate or severe flare according to the modified Safety of Estrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA SLEDAI) SLE Flare Index (modified excluded severe flares from the SELENA SLEDAI flare assessment that were triggered only by an increase in SLEDAI SLEDAI score to >12). Change in SELENA SLEDAI instrument score of greater than 12.
Part A: Percentage of Participants Achieving a ≥ 50% Improvement in Cutaneous Lupus Disease Area and Severity Index (CLASI) Activity Score at Week 52 | At Week 52
  CLASI is used to assess the cutaneous lesions of SLE. The CLASI activity score measures the inflammatory activity of the disease. The activity score evaluates erythema, scale/hypertrophy, mucous membrane lesions, recent hair loss, and non-scarring alopecia, measured at 13 anatomical sites on the skin. The total activity score ranges from 0 to 70. Higher scores indicate greater disease activity and severity in SLE.
Part A: Change from Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) -Fatigue at Week 52 | Baseline (Day 1) and at Week 52
  The FACIT-Fatigue is a 13-item participant-completed questionnaire used to assess the impact of fatigue over the previous 7 days. Item responses range from 0 (Not at All) to 4 (Very Much). The FACIT-Fatigue is scored as the sum of item responses, with range from 0 to 52, where higher scores indicate less fatigue and a better quality of life.
Part A: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), and AEs of Special Interest (AESIs) up to Week 52 | Up to Week 52
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in a participant's offspring; abnormal pregnancy outcomes; is a suspected transmission of any infectious agent via an authorized medicinal product; or other situations as per the Investigator's medical or scientific judgment. AESIs will include hypersensitivity or post-injection systemic reactions, infections of special interest, malignancy, psychiatric events, and fatal events.
Part B: Percentage of Participants Achieving Definition of Remission in SLE (DORIS) Remission at Week 104 | At Week 104
  DORIS remission is defined as clinical SLEDAI-2K equal to (=) 0 (excluding anti- double stranded deoxyribonucleic acid [dsDNA] and complement); and PGA less than (<) 0.5; and prednisone (or equivalent dose) < 5 mg/day on stable anti-malarial (AM), immunosuppressants (ISs) and biologic therapy.
Part B: Percentage of Participants Maintaining Systematic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SDI) of 0 up to Week 156 | Up to Week 156
  The SDI measures irreversible changes occurring since the diagnosis of SLE. The questionnaire contains 39 items covering 12 different organ systems. Individual ranges for organ systems are ocular: 0-2, neuropsychiatric: 0-6; renal: 0-3; pulmonary: 0-5; cardiovascular: 0-6; peripheral vascular: 0-5; gastrointestinal: 0-5; musculoskeletal: 0-6; skin: 0-3; endocrine (diabetes): 0-1; gonadal: 0-1; and malignancies: 0-2. The SDI score is calculated by summing the individual scores for 12 organ systems and ranges from 0 (no damage) to 45 (increasing disease damage) where higher score indicates increasing disease damage severity.
Part B: Number of Participants With AEs, SAEs, and AESIs up to Week 104 and Week 156 | Up to Week 104 and Week 156
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in a participant's offspring; abnormal pregnancy outcomes; is a suspected transmission of any infectious agent via an authorized medicinal product; or other situations as per the Investigator's medical or scientific judgment. AESIs will include hypersensitivity or post-injection systemic reactions, infections of special interest, malignancy, psychiatric events, and fatal events.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (104):
- United States (45):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Flagstaff, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Covina, California
  - GSK Investigational Site, Fontana, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Hills, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Temecula, California
  - GSK Investigational Site, Tujunga, California
  - GSK Investigational Site, Van Nuys, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Sugar Hill, Georgia
  - GSK Investigational Site, Morton Grove, Illinois
  - GSK Investigational Site, Rockford, Illinois
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Sparta, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Baytown, Texas
  - GSK Investigational Site, Colleyville, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Glendale, Wisconsin
- Argentina (9):
  - GSK Investigational Site, Berazategui
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Mar del Plata
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
- Brazil (8):
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Cuiabá
  - GSK Investigational Site, Juiz de Fora
  - GSK Investigational Site, Passo Fundo
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São José do Rio Preto
  - GSK Investigational Site, São Paulo
- France (6):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Toulouse
- Germany (4):
  - GSK Investigational Site, Herne
  - GSK Investigational Site, Lübeck
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Meerbusch
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion
  - GSK Investigational Site, Thessaloniki
- Italy (7):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Ferrara
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Reggio Emilia
  - GSK Investigational Site, Rome
  - GSK Investigational Site, Rozzano
- Japan (5):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Mexico (9):
  - GSK Investigational Site, Cuauhtémoc, Mexico City
  - GSK Investigational Site, DF
  - GSK Investigational Site, Guadalajara Jalisco
  - GSK Investigational Site, León
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Monterrey Nuevo LeOn
  - GSK Investigational Site, San Luis Potosí City
  - GSK Investigational Site, Torreón
- GSK Investigational Site, Almada, Portugal
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, VigoPontevedra
  - GSK Investigational Site, Villajoyosa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/